CLINICAL TRIAL: NCT02802826
Title: The Effects of a Tailored, Home-based Exercise Prescription to Increase Physical Activity in Breast Cancer Patients Undergoing Systemic Chemotherapy
Brief Title: Studying Tailored Exercise Prescriptions in Breast Cancer Patients
Acronym: STEPS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Dr Stephen Kihara, Chief Investigator, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Awaited
Record Dates: First submitted 2016-05-23; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Exercise; Chemotherapy; Physical Activity; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored Exercise Prescription (Experimental): Participants will have a discussion on the 'My Exercise Prescription' booklet on the benefits of increasing levels of physical activity. They will be encouraged to read this in more detail and guided through its completion. The participant will receive an exercise prescription using the Pre-Intervention Assessment Tool (PIAT) and following discussion with the participant on a realistic and achievable starting point.
  The booklets provided will guide participants through the exercise programme which is a graduated walking-based activity intervention. Both booklets provide participants with a suggested starting point for walking distance per week based on their PIAT score as well as motivational and behaviour change strategies to encourage participation.
  Interventions: Behavioral: Tailored Exercise Prescription
- Standard Care (No Intervention): No sham or placebo conditions will be used in the study. At visit 1 standard care participants will be given the Standard Care Information Sheet and asked to simply continue with standard care.

INTERVENTIONS:
Behavioral: Tailored Exercise Prescription — The intervention is a walking- based exercise prescription with the aim of a graduated increase in exercise to achieve national guidelines (i.e. Over 150mins of moderate intensity exercise over a week).
  Arms: Tailored Exercise Prescription

SUMMARY:
Chemotherapy forms a significant part of many breast cancer patient's treatment and is associated with various common, known adverse effects. For the last few decades, physical activity has been emerging as a viable intervention to help many of these adverse effects. The study will determine if the provision of a 12-week tailored walking programme, provided alongside a home-based exercise prescription from a cancer doctor results in improved levels of physical activity and quality of life in patients with breast cancer undergoing chemotherapy.

DETAILED DESCRIPTION:
Background Breast cancer is the most common cancer in females, with over 85% of women surviving their disease for 5 years or more. Chemotherapy forms a significant part of many patient's treatment and is associated with various common, well-characterised adverse effects. For the last few decades, physical activity has been emerging as a viable intervention to help many of the adverse effects of chemotherapy. Studies looking at patient's preferences have shown that the majority preferred walking, moderate-intensity, home-based exercise. Previous small studies have shown that cancer doctors have considerable influence on exercise behaviour; a simple recommendation significantly increased the activity levels of newly diagnosed breast cancer patients commencing treatment. A further question in the study will also assess the effect of exercise on markers of chronic inflammation in the blood. Exercise is known to reduce inflammation and this may play a significant role in cancer.

Method The study will determine if the provision of a 12-week tailored walking programme, provided alongside a home-based exercise prescription from a cancer doctor results in improved levels of physical activity in patients with breast cancer undergoing chemotherapy. Secondary objectives will assess patient-reported activity, quality-of-life, completion rates of chemotherapy, cognitive function, anxiety and depression levels, body composition as well as exploring the role of the effects on specific markers of chronic inflammation in the blood.

The investigators will recruit 100 patients from LRI undergoing chemotherapy for breast cancer. Participants will be allocated to either the intervention or a standard care group in this study. Those in the intervention group will receive the walking programme with various motivational strategies incorporated as well as a discussion on the benefits of exercise and a prescription from the cancer team. Those in the standard care will not receive the intervention material. All women will wear wrist accelerometers (to measure activity levels) before and after the 12-week period and complete assessments at these points (as well as a further follow up assessment at 6 months). Assessments will include study questionnaires, cognitive testing, measurements of body fat and blood tests.

Potential impact The investigators aim to show that the intervention will result in significantly improved levels of physical activity, as well as improved quality of life and improvements in other secondary outcome measures. They also predict that the intervention will result in a significant lowering of inflammatory marker concentration when compared to standard care. The study will provide an important addition to the evidence that exists for cancer teams to encourage patients and survivors to meet national physical activity guidelines. In the longer term, the intervention being tested in the proposed study has the potential to be an inexpensive and sustainable addition to the standard care provided to cancer patients and this will hopefully lead to a larger-scale national study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to admission to the study.
* Age 18-75 years of age.
* Able to read and speak English.
* Not currently meeting national guidelines for exercise (i.e. <150mins moderate intensity exercise on 5 or more days per week).
* Histologically confirmed diagnosis of primary breast malignancy (GROUP 1), OR Histological or radiological confirmation of advanced/metastatic breast malignancy (GROUP 2).
* Due to commence (or within 3 weeks of commencing) neo-adjuvant or adjuvant systemic chemotherapy for breast malignancy (GROUP 1), OR Due to commence (or within 3 weeks of commencing) any line of palliative systemic chemotherapy for breast malignancy (GROUP 2).
* ECOG Performance Status 0-2.
* Able (in investigator's opinion) to be able to comply with all study requirements and exercise prescription.

Exclusion Criteria:

* Any severe or uncontrolled medical conditions.
* Any unstable or uncontrolled cardiopulmonary illness.
* Recent Myocardial Infarction (<6months)
* Implanted Cardiac defibrillator.
* Uncontrolled Hypertension
* Pregnancy or <12 weeks post-partum.
* Life expectancy <3 months.
* Prior history of neurological or psychiatric disorder, which could cause cognitive deficits.
* Current or planned enrolment in structured exercise or weight loss programme.
* Injury, disability or symptoms preventing compliance with exercise prescription.
* Psychological, sociological or geographical conditions that do not permit compliance with the study protocol or exercise prescription.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Level of Moderate-Vigorous Physical Activity | A Change between baseline and 3 months (post intervention)
  To determine whether tailored home-based exercise prescriptions results in a change in Physical Activity (objectively measured) in patients with breast cancer undergoing systemic chemotherapy. Measured by accelerometer.

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQOL) | A Change between baseline, 3 months (post intervention), and 6 months.
  Does the intervention result in improved HRQOL in patients undergoing systemic chemotherapy. Measured by Euro-QOL 5D.
Health-Related Quality of Life (HRQOL) 2 | A Change between baseline, 3 months (post intervention), and 6 months.
  Does the intervention result in improved HRQOL in patients undergoing systemic chemotherapy. Measured by EORTC QLQ C30.
Subjectively measured physical activity | A Change between baseline, 3 months (post intervention), and 6 months.
  Does the intervention result in improved Subjectively measured physical activity in patients undergoing systemic chemotherapy. Measured by International Physical Activity Questionnaire.
Sitting time | Baseline, 3 months (post intervention) & 6 months
  Does the intervention result in improved sitting time in patients undergoing systemic chemotherapy. Measured by International Physical Activity Questionnaire.
Alteration in Stage of Motivational Readiness to Change | A Change between baseline, 3 months (post intervention), and 6 months.
  Does the intervention result in improved Stage of Motivational Readiness to Change in patients undergoing systemic chemotherapy. Measured by Stages of Change Questionnaire.
Completion rate of Systemic Chemotherapy | 6 months.
  Does the intervention result in improved chemotherapy completion in patients undergoing systemic chemotherapy. Measured by data collected on completion rate of chemotherapy.
Subjective Cognitive Function | A Change between baseline, 3 months (post intervention), and 6 months.
  Does the intervention result in improved subjective cognitive function in patients undergoing systemic chemotherapy. Measured by Cognitive Failures Questionnaire.
Objective Cognitive Function | A Change between baseline, 3 months (post intervention), and 6 months.
  Does the intervention result in improved objective cognitive function in patients undergoing systemic chemotherapy. Measured by objective cognitive testing.
Body Composition | A Change between baseline, 3 months (post intervention), and 6 months.
  Does the intervention result in favourable changes in body composition with an increase in lean body mass (LBM) and a reduction in body fat percentage (BFP) in patients undergoing systemic chemotherapy. Measured by Bioelectrical Impedance Analysis.

OTHER OUTCOMES:
To explore whether the tailored home-based exercise prescription has an effect on the concentration of circulating markers of low-grade chronic inflammation (1) | A Change between baseline and 3 months (post intervention)
  Measured plasma levels of IL-6. Measures at baseline and post-intervention.
To explore whether the tailored home-based exercise prescription has an effect on the concentration of circulating markers of low-grade chronic inflammation (2) | A Change between baseline and 3 months (post intervention)
  Measured plasma levels of TNF-alpha. Measures at baseline and post-intervention.
To explore whether the tailored home-based exercise prescription has an effect on the concentration of circulating markers of low-grade chronic inflammation (3) | A Change between baseline and 3 months (post intervention)
  Measured plasma levels of CRP. Measures at baseline and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kihara, MBChB MRCP, Study Chair — University of Leicester NHS Trust
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No